CLINICAL TRIAL: NCT04714346
Title: Effects of Trendelenburg Position and Pneumoperitonium on Cerebral Tissue Oxygen Saturation and Early Postoperative Cognitive Dysfunction (POCD) in Patients Undergoing Laparoscopic Major Abdominal Oncological Surgery
Brief Title: Does Positioning Effects on Early Postoperative Cognitive Dysfunction in Laparoscopic Oncological Surgery
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, hazal ozkaya hız, Effects of Trendelenburg position and pneumoperitonium on cerebral tissue oxygen saturation and early postoperative cognitive dysfunction (POCD) in patients undergoing laparoscopic major abdominal oncological surgery, Saglik Bilimleri Universitesi
Other Study IDs: 2019-08/384
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Ischemic Attack, Transient
Keywords: POCD; Trendelenburg position; pneumoperitonium; NIRS; MMSE
MeSH Terms: conditions — Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: no interventions — there is no intervention

SUMMARY:
Laparoscopic surgery is an alternative to open surgical techniques for reasons such as less blood loss,less need for transfusion, shorter discharge time. In laparoscopic cases, various positions are given to patients, especially trendelenburg, in order to remove organs and see the area of the operation more easily. The Trendelenburg position causes cerebrovascular changes.Several studies have reported an increase in intracranial pressure (ICP)at the Trendelenburg position. There are also studies that show brain tissue oxygen saturation (SctO2) decreases in this position. Research has reported that cerebral perfusion pressure decreases if the position lasts longer.When pneumoperitonium is administered during laparoscopic surgery, cerebral blood flow may increase as a result of the increase in PaCO2.Brain tissue oxygen saturation depends on blood flow.There is also an inverse ratio between end tidal CO2. To prevent deterioration of cerebral function, methods are needed that determine the onset of desaturation and make early intervention possible.

The method,known as near-infrared spectroscopy (NIRS), offers a fixed non-invasive and safe method of determining cerebral desaturation.In addition, NIRS has the potential to improve patient outcomes, reduce postoperative complications and duration of post-anesthesia care.Changes in NIRS measurement values associated with position, especially today, are seen in cerebral perfusion in patients undergoing major surgery, oxygenation and postop have been associated with cognitive dysfunction in the process.Postoperative cognitive dysfunction is associated with increased mortality and therefore it is very important to identify factors that increase risk in order to take appropriate protective measures.Intracerebral ischemia and desaturation may be responsible for the development of POCD.

In this study, we aimed to observe NIRS changes due to Trendelenburg position and pneumoperitonium in patients undergoing laparoscopic major abdominal oncological surgery and to examine the effect of POCD on early stage.

DETAILED DESCRIPTION:
In Saglık Bilimleri University, Ankara A.Y. Oncology Research and Trainnee Hospital, Anesthesiology and reanimation clinic,patients who are scheduled for elective laparoscopic major abdominal surgery after the approval of the Ethics Committee will be enrolled in the study. From the beginning of the study, successive patients were included in the study. Measurement values were taken and recorded using the NIRS device in our clinic throughout the case in patients 18 years of age and older. All patients were evaluated with MMSE in preoperative and postoperative period. According to power analysis using mean and standard deviation to determine the sample size of the patients to be taken in this process, at least 52 patients were planned to be included in the study.

After preoperative MMSE testing, ASA scores, comorbidities,demographic data, drugs used in anesthesia, vasopressor use, pneumoperitonium pressures and duration, angle and duration of trendelenburg position, and vital parameters were recorded with NIRS device in our clinic.

MMSE test was re-administered to all patients in the first week of postoperative period.

Patients with preoperative MMSE score (M0) 24/30 points and above; postoperative 7th day (M1) was re-evaluated and those with a fall of 4 points and more in M1 score than M0 score were assessed as POCD.

NIRS measurements were taken perioperative and their correlation with POCD was looked at.

Inclusion criteria;

* 18 years and older,
* preoperative 24 points and above on MMSE test(M0)
* Laparoscopic major abdominal oncological surgery planned patients who will receive general anesthesia.

Exclusion criteria;

* People with a history of cerebral ischemia or hemorrhage,
* Those with a history of neurodegenerative disease,
* Those with diagnosed carotid stenosis,
* Those with a score of 23 and below on the MMSE test,
* Those with a history of Carotid Endarterectomy,
* Patients who have undergone aneurysm surgery,
* Those who are addicted to alcohol,
* Those with psychiatric illness,
* Those who have undergone cervical surgery,
* Those with a history of transient ischemic attacks,

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above,
* 24 points and above on MMSE test,
* Laparoscopic major abdominal oncological surgery planned patients who will receive general anesthesia

Exclusion Criteria:

* People with a history of cerebral ischemia or hemorrhage,
* Those with a history of neurodegenerative disease,
* Those with diagnosed carotid stenosis,
* Those with a score of 23 and below on the MMSE test,
* Those with a history of Carotid Endarterectomy,
* Patients who have undergone aneurysm surgery,
* Those who are addicted to alcohol,
* Those with psychiatric illness,
* Those who have undergone cervical surgery,
* Those with a history of transient ischemic attacks,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who do not meet the exclusion criteria will undergo laparoscopic major abdominal oncological surgery over the age of 18.
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
MMSE changings in POCD | each patient in seven days
  Lowest MMSE score is 0;highest is 30. 24 is the limit of mild cognitive decline. In MMSE, to evaluate cognitive changings 4 point of decline is meaningful. Primarily, In our study, First patients with preoperative MMSE score(M0) 24/30 points and above will be re-evaluated on postoperative seventh day(M1) and those with a decrease of 4 points and greater than M0 score in M1 score will be evaluated as POCD.

SECONDARY OUTCOMES:
NIRS measurement correlation | each patient in seven days
  NIRS value of rSO2 changings was looked at. Rate of %20 and above were recorded as meaningful.
  Secondarily, NIRS measurements will be taken perioperative and their correlation with POCD will be looked at.

CONTACTS AND LOCATIONS:
Locations (1):
- SBU. Ankara A.Y. Oncology Research and Training Hospital, Ankara, Turkey (Türkiye)